CLINICAL TRIAL: NCT02970292
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Adjunctive Pimavanserin for the Treatment of Schizophrenia
Brief Title: Efficacy and Safety of Adjunctive Pimavanserin for the Treatment of Schizophrenia (ENHANCE-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-034; 2016-003434-24 (EudraCT Number)
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pimavanserin (Experimental): Drug- pimavanserin 34 mg, 20 mg, or 10 mg taken as two tablets + background antipsychotic, once daily by mouth
  Interventions: Drug: Pimavanserin
- Placebo (Placebo Comparator): Placebo + background antipsychotic, taken as two tablets, once daily by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg, 20 mg, or 10 mg , taken as two tablets once daily by mouth
  Arms: Pimavanserin
Drug: Placebo — Placebo, taken as two tablets, once daily by mouth
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of adjunctive pimavanserin compared with adjunctive placebo in the treatment of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

1. Adults patients, between 18 and 55 years of age
2. A clinical diagnosis of schizophrenia with a minimum duration of 1 year
3. The main background antipsychotic with which the subject is being treated must be one of the antipsychotics listed below:

   * Aripiprazole
   * Aripiprazole long-acting injectables:

     * Abilify Maintena®
     * Aristada®
   * Risperidone
   * Risperidone long-acting injection
   * Olanzapine
   * Lurasidone
   * Cariprazine
   * Brexpiprazole
   * Asenapine
4. Has had a partial but inadequate response to antipsychotic treatment
5. Has a history of response to antipsychotic treatment other than clozapine

Exclusion Criteria:

1. Patient has a psychiatric disorder other than schizophrenia
2. Patient has a history of resistance to antipsychotic treatment
3. A urine drug screen (UDS) result at Baseline that indicates the presence of any tested prohibited substance of potential abuse, except marijuana

   a. Patients with a result indicating the presence of marijuana are permitted if they agree to abstain from marijuana use during the study and the medical monitor approves the subject's participation
4. Patient has current evidence of a serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies, which would affect the patient's ability to participate in the program
5. Patient has had a myocardial infarction in the last six months
6. Patient is taking a medication or drug that prolongs the QT interval or has a family or personal history or symptoms of long QT syndrome

Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (82):
- United States (30):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Rogers, Arkansas
  - Bellflower, California
  - Cerritos, California
  - Culver City, California
  - Lemon Grove, California
  - Long Beach, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Boca Raton, Florida
  - Lauderhill, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Lake Charles, Louisiana
  - Catonsville, Maryland
  - Ann Arbor, Michigan
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Cedarhurst, New York
  - Jamaica, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Dayton, Ohio
  - Charleston, South Carolina
  - Richardson, Texas
  - Salt Lake City, Utah
- Bulgaria (9):
  - Burgas
  - Pazardzhik
  - Plovdiv
  - Sofia
  - Targovishte
  - Tserova Koria
  - Varna
  - Veliko Tarnovo
  - Vratsa
- Canada (3):
  - Chatham, Ontario
  - Montreal, Quebec
  - Toronto
- Czechia (4):
  - Hradec Králové
  - Pilsen
  - Prague
  - Říčany
- Hungary (4):
  - Kalocsa, Bács-Kiskun Megya
  - Budapest, Pest County
  - Debrecen
  - Pécs
- Lithuania (3):
  - Kaunas
  - Šilutė
  - Vilnius
- Poland (4):
  - Bialystok
  - Bydgoszcz
  - Lublin
  - Pruszcz Gdański
- Russia (11):
  - Roshchino, Leningradskaya Oblast'
  - Plekhanovo, Lipetsk Oblast
  - Tonnel’nyy, Stavropol Kray
  - Arkhangelsk
  - Moscow
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
  - Voronezh
  - Yaroslavl
- Serbia (4):
  - Belgrade
  - Kovin
  - Kragujevac
  - Niš
- Ukraine (10):
  - Kherson, Vil. Stepanivka
  - Dnipro
  - Hlevakha
  - Kharkiv
  - Kyiv
  - Odesa
  - Oleksandrivka
  - Poltava
  - Smila
  - Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bugarski-Kirola D, Abbs B, Odetalla R, Liu IY, Darwish M, DeKarske D. Adherence to Background Antipsychotic and Pimavanserin in Patients with Schizophrenia: Post Hoc Analyses from the ENHANCE and ADVANCE Studies. Patient Prefer Adherence. 2024 Jan 19;18:207-216. doi: 10.2147/PPA.S436041. eCollection 2024. PMID 38264323

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimavanserin: Patients started treatment with pimavanserin 20 mg once daily (QD). At the Week 1, Week 2 and Week 3 visit, the dose could be increased to 34 mg QD or decreased to 10 mg QD at the investigator's discretion (to improve symptom reliev or tolerability, respectively). Thereafter, the daily dose was to remain the same for the remainder of the study.
  Patients were to continue their background antipsychotic treatment.
- Placebo: Pimavanserin-matching Placebo.
  Patients were to continue their background antipsychotic treatment.
Period: Overall Study
Arm/Group | Pimavanserin | Placebo
Started | 198 | 198
Completed | 174 | 190
Not Completed | 24 | 8
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Noncompliance with study drug | 2 | 2
Not completed — Adverse Event | 5 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomised and treated with at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimavanserin | Placebo | Total
Number analyzed (Participants) | 198 | 198 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (9.42) | 37.4 (9.45) | 37.1 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 78 | 150
  Male | 126 | 120 | 246
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 22 | 44
  White | 176 | 172 | 348
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 2 | 2
  Hungary | 3 | 3 | 6
  United States | 37 | 34 | 71
  Czechia | 1 | 1 | 2
  Ukraine | 16 | 24 | 40
  Poland | 3 | 3 | 6
  Bulgaria | 43 | 50 | 93
  Lithuania | 3 | 6 | 9
  Serbia | 44 | 33 | 77
  Russia | 48 | 42 | 90
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.74 (4.177) | 26.92 (4.029) | 26.83 (4.099)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a 30-item scale used to evaluate the presence, absence, and severity of schizophrenia symptoms. The 30 items are arranged as 7 positive symptom items (P1 to P7), 7 negative symptom items (N1 to N7), and 16 general psychopathology symptom items (G1 to G16). Items are scored over the past week (7 days) on a 7-point scale ranging from 1 (absent) to 7 (extreme). The PANSS total score can range from a minimum of 30 to a maximum of 210, where a higher score signifies greater severity of schizophrenia symptoms.
Time Frame: From baseline to Week 6
Population: Patients randomised and treated (at least 1 dose of study medication) who had both a baseline value and at least 1 post-baseline value for the PANSS total score.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
score on a scale
  Baseline | 88.3 (0.68) | 88.1 (0.61)
  Change from baseline to Week 6: number analyzed (Participants) | 173 | 189
  Change from baseline to Week 6 | -15.3 (0.93) | -13.4 (0.83)
Statistical Analysis 1: Comparison: Pimavanserin vs Placebo; Test type: Superiority; p = 0.0940, mixed-effects model for repeated measure; Difference in MMRM LSMs = -2.1, 95% CI 2-sided [-4.5 to 0.4], Standard Error of Mean 1.24

2. Secondary Outcome: Change From Baseline to Week 6 in the Clinical Global Impression-Severity (CGI-S) Score
Description: The CGI-S is a 1-item scale, used to rate the severity of the disorder from 0 (not assessed) to 7 (among the most extremely ill patients). A higher CGI-S score denotes greater severity of the disorder.
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
score on a scale
  Baseline | 4.6 (0.04) | 4.6 (0.04)
  Change from baseline to Week 6: number analyzed (Participants) | 173 | 189
  Change from baseline to Week 6 | -0.8 (0.06) | -0.7 (0.05)

3. Secondary Outcome: Change From Baseline (CFBL) to Week 6 in PANSS Subscale Scores, i.e. PANSS Positive Subscale Score, PANSS Negative Subscale Score and PANSS General Psychopathological Scale Score
Description: The PANSS is a 30-item scale used to evaluate the presence, absence, and severity of schizophrenia symptoms. The 30 items are arranged as 7 positive symptom items (P1 to P7), 7 negative symptom items (N1 to N7), and 16 general psychopathology symptom items (G1 to G16). Items are scored over the past week (7 days) on a 7-point scale ranging from 1 (absent) to 7 (extreme).
  The PANSS positive subscale score can range from 7 to 49; the PANSS negative subscale score can range from 7 to 49; the PANSS general psychopathology scale score can range from 16 to 112.
  For each of the subscale scores, a higher score signifies greater severity of schizophrenia symptoms.
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
score on a scale
  PANSS positive scale BL | 23.0 (0.25) | 22.8 (0.23)
  PANSS positive scale CFBL to 6 weeks: number analyzed (Participants) | 173 | 189
  PANSS positive scale CFBL to 6 weeks | -5.4 (0.34) | -4.9 (0.30)
  PANSS negative scale BL | 23.0 (0.29) | 23.1 (0.29)
  PANSS negative scale CFBL to 6 weeks: number analyzed (Participants) | 173 | 189
  PANSS negative scale CFBL to 6 weeks | -2.8 (0.28) | -2.1 (0.28)
  PANSS general psychopatholigy scale BL | 42.4 (0.45) | 42.2 (0.45)
  PANSS gen. psychopath. scale CFBL to 6 w: number analyzed (Participants) | 173 | 189
  PANSS gen. psychopath. scale CFBL to 6 w | -7.2 (0.47) | -6.4 (0.47)

4. Secondary Outcome: PANSS Responders
Description: Porportion of patients showing a PANSS response of >=20% or >=30% reduction in PANSS total score PANSS total score reduction signifies improvement.
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
Participants
  PANSS total score reduction >=20% | 109 | 99
  PANSS total score reduction >=30% | 71 | 67

5. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Response
Description: The CGI-I is a 1-item scale, used to rate the improvement from 1 (very much improved) to 7 (very much worse). Higher scores denote less improvement.
  A CGI-I score of 1 or 2 was counted as response. The Analysis was performed twice; once including missing values as non-responders (MN) and once including only observed cases (OC).
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
Participants
  CGI-I response (MN) | 68 | 65
  CGI-I response (OC): number analyzed (Participants) | 173 | 189
  CGI-I response (OC) | 68 | 65

6. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at Week 6
Description: The CGI-I is a 1-item scale, used to rate the improvement from 1 (very much improved) to 7 (very much worse). Higher scores denote less improvement.
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 173 | 189
score on a scale | 2.8 (0.07) | 3.0 (0.07)

7. Secondary Outcome: Change From Baseline to Week 6 in Personal and Social Performance (PSP) Scale Score
Description: The PSP is a validated 100-point (1 to100) single-item rating scale to assess the psychosocial functioning of patients with schizophrenia. The maximum score is 100. Higher scores denote better psychosocial functioning.
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
score on a scale
  Baseline | 51.8 (0.79) | 51.6 (0.78)
  Change from baseline to Week 6: number analyzed (Participants) | 173 | 188
  Change from baseline to Week 6 | 6.8 (0.71) | 5.7 (0.64)

8. Secondary Outcome: Drug Attitude Inventory (DAI-10)
Description: The DAI-10 contains 6 items (1, 3, 4, 7, 9, and 10) that a patient who is fully adherent to study medication would answer as "True" and 4 items (2, 5, 6, and 8) that a patient who is fully adherent to study medication would answer as "False." A correct answer is scored +1 and an incorrect answer is scored -1; the total score is derived as overall sum. The score can range from -10 to 10. Positive total scores indicate adherence and negative total scores indicate non-adherence. Higher scores denote better adherence.
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
score on a scale
  Baseline | 5.6 (0.24) | 5.8 (0.23)
  Change from baseline to Week 6: number analyzed (Participants) | 173 | 188
  Change from baseline to Week 6 | 0.4 (0.20) | 0.4 (0.20)

9. Secondary Outcome: Change From Baseline to Week 6 in Karolinska Sleepiness Scale (KSS) Score
Description: The KSS is a self-reported measure of a patient's level of drowsiness. In this study, drowsiness was to be rated during the last week (7 days). Scoring is based on a 9-point verbally anchored scale ranging from 1 (extremely alert) to 9 (very sleepy, great effort to keep awake, fighting sleep). The maximum score is 9. Higher scores denote more drowsiness.
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 193 | 196
score on a scale
  Baseline | 4.6 (0.11) | 4.7 (0.12)
  Change from baseline to Week 6: number analyzed (Participants) | 173 | 189
  Change from baseline to Week 6 | -0.5 (0.12) | -0.2 (0.12)

ADVERSE EVENTS:
Time Frame: From baseline to Week 6
Description: The analysis population were those patients who received at least one dose of the study drug. Patients were classified according to the actual treatment received.
Arm/Group | Pimavanserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/198
Serious Adverse Events (participants affected / at risk) | 2/198 | 2/198
Other Adverse Events (participants affected / at risk) | 31/198 | 31/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=198) | Placebo (N=198)
Schizophrenia (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucination auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=198) | Placebo (N=198)
Headache (Nervous system disorders) | 13 (16) | 18 (24)
Somnolence (Nervous system disorders) | 13 (19) | 7 (8)
Insomnia (Psychiatric disorders) | 10 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's Prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT02970292/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT02970292/SAP_001.pdf